CLINICAL TRIAL: NCT07201844
Title: ORIGAMI: Internetbaserad Behandling för GAD. Effekten av Att få välja Behandling själv Samtbehandlarens förmåga Att Matcha Patienter Till rätt Behandling. En Randomiserad kontrolleradprövning.
Brief Title: The Effect of Patient Preference for Treatment Model in Internet Delivered Cognitive Behavior Therapy for Generalized Anxiety Disorder
Acronym: ORIGAMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Forsell, Principal Researcher, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-03553-01 RCT2
Record Dates: First submitted 2025-09-16; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Generalized Anxiety Disorder (GAD)
Keywords: Internet interventions; Digital mental health services; cognitive behaviour therapy; patient preferences; psychiatry
MeSH Terms: conditions — Generalized Anxiety Disorder; Patient Preference

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants who do not get to choose treatment are not aware that they could have been assigned to do so.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment choice (Experimental): Patients have been randomized to getting to read about and then choose one of the two treatments
  Interventions: Behavioral: Metacognitive Internet delivered Cognitive Behavior Therapy; Behavioral: Intolerance of uncertainty based Internet delivered Cognitive Behavior Therapy
- Random assignment to treatment (Experimental): Patients have been directly randomized into one of the two treatments
  Interventions: Behavioral: Metacognitive Internet delivered Cognitive Behavior Therapy; Behavioral: Intolerance of uncertainty based Internet delivered Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Metacognitive Internet delivered Cognitive Behavior Therapy — Specialist Guided Internet delivered Cognitive Behavior Therapy based on the metacognitive model of excessive worry
Behavioral: Intolerance of uncertainty based Internet delivered Cognitive Behavior Therapy — Specialist Guided Internet delivered Cognitive Behavior Therapy based on the Intolerance of uncertainty model of excessive worry

SUMMARY:
The goal of this clinical trial is to investigate the effect of allowing patients to choose between two internet-based cognitive behavioral treatments (ICBT) for generalized anxiety disorder (GAD). The goal is also to examine psychologists' ability to predict which of the two treatments the patient will benefit most from.

The main questions it aims to answer are:

* Do patients who are randomized to choose their treatment improve more in their GAD symptoms compared to patients who are randomly assigned to a treatment?
* Does allowing patients to choose their treatment increase treatment adherence, compared to being randomly assigned to a treatment?
* Does allowing patients to choose their treatment increase treatment satisfaction and credibility, compared to being randomly assigned to a treatment?
* Does allowing patients to choose their treatment increase patients' sense of agency related to the treatment process, compared to being randomly assigned to a treatment?
* Do patients who receive a treatment that matches the psychologist's prediction of which treatment would fit the patient best show better treatment outcomes (primarily reduction in GAD symptoms over time, but also secondary outcomes such as satisfaction), compared to patients who receive a treatment that does not match the psychologist's prediction?

Participants included in the trial will be randomized to one of two conditions: 1) read short descriptions of the two treatment programs and based on that choose the preferred treatment, 2) randomly being allocated to one of the two treatments. The two internet-based treatment programs which the patients can choose between or be randomly allocated to are: 1) Intolerance of uncertainty-based ICBT and 2) Metacognition-based ICBT. Both programs consist of 8 treatment modules and run for 10 weeks. Patients in both conditions receive continuous support by a psychologist through a built-in message function on the treatment platform. The patient will receive feedback from the psychologist on their assignments and exercises and the psychologist will respond to the participants' messages.

DETAILED DESCRIPTION:
A randomized trial will be conducted within the Internet Psychiatry Clinic in Stockholm. An option will be added to the online sign-up form giving potential patients the option to participate in a treatment for GAD as part of this study. Based on information provided in the sign-up-form and an assessment via video-call with a psychologist, patients will be included/excluded.

Included patients will be randomized (2:1:1) to either 1) read short descriptions of the two treatment programs and based on that choose the preferred treatment or 2) being randomly assigned to one of the two treatments. In both conditions, a psychologist will make a prediction regarding which of the two treatments the patient will benefit most from, based on their clinical assessment of the patient. The treatment effect for patients who were either randomly assigned to, or chose, a treatment that matches the psychologist's prediction will be compared with the treatment effect for patients who were either randomly assigned to, or chose, a treatment that does not match the psychologist's prediction.

The two internet-based treatment programs which the patients can choose between or be randomly allocated to are: 1) Intolerance of uncertainty-based ICBT and 2) Metacognition-based ICBT. These programs will be conducted as part of regular care at the Internet Psychiatry Clinic in Stockholm, meaning that each patient will undergo the regular assessment process at the clinic. Both programs are ICBT programs of similar scope, consisting of 8 modules to be completed during 10 weeks. During this time patients read written material which instructs them to do specific exercises and answer specific questions. The patient can message a psychologist at the clinic via a built-in message function on the treatment platform.

Primary outcome to assess treatment effect in this study is change in GAD-symptoms (measured with GAD-7) from pre-treatment to post-treatment. Secondary outcome measures to assess treatment effect is patients' satisfaction with the treatment program post-treatment (measured with Client satisfaction questionnaire), how credible the patient consider the treatment program to be (measured with Treatment Credibility Questionnaire 2 weeks after treatment start) and patients' sense of agency related to their treatment process (measured with Therapeutic Agency Inventory 4 weeks after treatment start). Patients' adherence to the treatment program will be assessed by the number of completed modules by the end of treatment.

A power analysis has shown that n=200 in each arm gives at least 80% power to detect a minimally clinically significant effect of d=.24. Based on similar treatments at the Internet Psychiatry Clinic the investigators expect around 10% drop-out meaning that the aim is to include 440 patients in total to get 200 in each arm.

Hypothesis 1: Patients who are allowed to choose their preferred treatment will exhibit a greater treatment effect (specified above) compared to patients who are randomly assigned to a treatment.

Hypothesis 2: Patients will 1) have a higher sense of agency in their treatment process, 2) be more satisfied with the treatment, 3) be more adherent to the treatment and 4) will rate the treatment as more credible if they themselves get to choose treatment compared to random assignment.

Hypothesis 3: Patients who receive a treatment that matches the psychologist's prediction will exhibit a greater treatment effect (specified above), compared to patients who receive a treatment that does not match the psychologist's prediction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Meet diagnostic criteria for GAD according to DSM-5, as assessed by a psychologist on a video-call.
* Self-rated score ≥ 7 on GAD-7.
* Can read and speak Swedish fluently.
* Have access to a smartphone, tablet, or computer and a Swedish BankID which allows access to the video-calls and treatment platform.
* Have the time and possibility to participate in the 10 week treatment.
* Consents to participate.

Exclusion Criteria:

* Patients that are judged to be in greater need of another psychiatric treatment for another psychiatric diagnosis (for example severe depression) and/or is judged to have a high risk of suicide.
* Current drug or alcohol abuse.
* Current severe somatic health concern or social vulnerability if this is judged to be too great an obstacle for the patient to carry out the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Generalized Anxiety Disorder - score (GAD-7) | Measured weakly from treatment start (pre-treatment) to 10 weeks after treatment start (post-treatment).
  Measures generalized anxiety symptoms. 7 items. Scores range from 0-21 with higher scores indicating more generalized anxiety

SECONDARY OUTCOMES:
Therapeutic Agency Inventory (adapted to the clinic) | 4 weeks after treatment start.
  Measures patients' sense of agency related to their treatment process. 15 items. Scores range from 0-75 with higher scores indicating a higher degree of agency.
Penn-State Worry Questionnaire (PSWQ) | At start of treatment (pre-treatment) and at 10 weeks after treatment start (post-treatment).
  Measures trait worry. 16 items. Scores range from 16-80 with higher scores indicating more worry.
Client satisfaction questionnaire (adapted to the clinic) | 10 weeks after treatment start (post-treatment).
  Measures satisfaction with treatment. 8 items. Scores range from 8-32 with higher scores indicating more satisfaction with the treatment.
Treatment Credibility Questionnaire (adapted to the clinic) | 2 weeks after treatment start.
  Measures treatment rationale credibility. 5 items. Scores range from 0-50 with higher scores indicating higher treatment credibility.
Montomery-Asberg Depression Rating Scale - Self-rated (MADRS-S) | Measured weakly from treatment start (pre-treatment) to 10 weeks after treatment start (post-treatment).
  Measures depression symptoms. 9 items. Scores range from 0 to 54 with higher scores indicating more depression symptoms.
Patient Health Questionnaire-9 (PHQ-9) | At start of treatment (pre-treatment) and at 10 weeks after treatment start (post-treatment).
  Measures depression symptoms. 9 items. Scores range from 0-27 with higher scores indicating more depressive symptoms.
World Health Organization Disability Assessment Schedule 2.0 | At start of treatment (pre-treatment) and at 10 weeks after treatment start (post-treatment).
  Measures disability/functional impairment. 12 items. Scores range from 0-48 with higher scores indicating a higher degree of impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Internet Psychiatry Clinic, Psychiatry Southwest, SLSO, Region Stockholm, Stockholm, Huddinge 14135, Stockholm, Sverige, Sweden

IPD SHARING:
Plan to Share IPD: No
All IPD will be confidential patient records and as such are not shareable.